CLINICAL TRIAL: NCT00024349
Title: 2X2 Factorial Randomized Phase III Study Comparing Standard Versus Reduced Volume Radiotherapy With and Without Synchronous Chemotherapy in Muscle Invasive Bladder Cancer
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With Stage II or Stage III Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068921; CRC-BC2001; EU-20052; ISRCTN68324339
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Fluorouracil; Mitomycin; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: mitomycin C
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy such as fluorouracil and mitomycin use different ways to stop tumor cells from dividing so they stop growing or die. Fluorouracil and mitomycin may make the tumor cells more sensitive to radiation therapy. It is not yet known if radiation therapy is more effective with or without chemotherapy in treating bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy to all or part of the bladder with or without chemotherapy in treating patients who have stage II or stage III bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of standard volume radiotherapy vs reduced volume radiotherapy with or without synchronous fluorouracil and mitomycin in patients with stage II or III (muscle invasive) bladder cancer.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, prior neoadjuvant chemotherapy (yes vs no), and intent to enter only 1 of the possible 2 randomizations on study (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo standard radiotherapy once daily 5 days a week for 4 or 6.5 weeks. Patients also receive synchronous chemotherapy comprising mitomycin IV on day 1 and fluorouracil IV continuously over days 1-5 and 16-20 during radiotherapy.
* Arm II: Patients undergo standard radiotherapy as in arm I (without chemotherapy).

If standard radiotherapy is clearly indicated (e.g., patients with multiple tumors) patients may be randomized to standard radiotherapy with or without chemotherapy (arms I or III above). If chemotherapy is clearly contraindicated, patients are randomized to standard or reduced volume radiotherapy without chemotherapy (arms III or IV above).

Quality of life is assessed at baseline, at the end of therapy, at 6 and 12 months post-randomization, and then annually for at least 5 years.

Patients are followed at 6, 9, and 12 months post-randomization and then at least annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive bladder cancer (T2-4a, N0, M0)

  * Adenocarcinoma
  * Transitional cell carcinoma
  * Squamous cell carcinoma
* Localized muscle invasion by surgery or imaging

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT or AST less than 1.5 times ULN

Renal:

* Glomerular filtration rate greater than 25 mL/min

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No inflammatory bowel disease
* No other prior malignancy within the past 2 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No other prior malignancy or uncontrolled systemic disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the pelvis

Surgery:

* See Disease Characteristics
* No bilateral hip replacements

Other:

* No concurrent metronidazole during fluorouracil administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2001-06; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Loco-regional disease free survival at 2 years

SECONDARY OUTCOMES:
Disease-free survival, metastases-free survival, and late toxicity by RTOG and Lent Som toxicity scores, Bladder capacity, and patient assessed Fact-BL quality of life scores at 1 and 2 years
Acute toxicity and cystoscopic local control at 3 months, 1 year, and 2 years
Rate of salvage cystectomy
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D. James, MD, Study Chair — University Hospital Birmingham
Locations (27):
- United Kingdom (27):
  - Royal United Hospital, Bath, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Royal Bournemouth Hospital NHS Trust, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - St. Thomas' Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Torbay Hospital, Torquay, England
  - Good Hope Hospital Trust, West Midlands, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Glan Clwyd Hospital, Rhyl, Wales

REFERENCES:
- [Result] James ND, Hussain SA, Hall E, Jenkins P, Tremlett J, Rawlings C, Crundwell M, Sizer B, Sreenivasan T, Hendron C, Lewis R, Waters R, Huddart RA; BC2001 Investigators. Radiotherapy with or without chemotherapy in muscle-invasive bladder cancer. N Engl J Med. 2012 Apr 19;366(16):1477-88. doi: 10.1056/NEJMoa1106106. PMID 22512481
- [Derived] Choudhury A, Porta N, Hall E, Song YP, Owen R, MacKay R, West CML, Lewis R, Hussain SA, James ND, Huddart R, Hoskin P; BC2001 and BCON investigators. Hypofractionated radiotherapy in locally advanced bladder cancer: an individual patient data meta-analysis of the BC2001 and BCON trials. Lancet Oncol. 2021 Feb;22(2):246-255. doi: 10.1016/S1470-2045(20)30607-0. PMID 33539743